CLINICAL TRIAL: NCT06189469
Title: Is Urdu Version of the King's Health Questionnaire a Reliable and Valid Tool
Brief Title: Reliability and Validity of Urdu Version of the King's Health Questionnaire
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC-FSD-00257
Record Dates: First submitted 2022-07-24; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Urinary Incontinence
Keywords: Urinary Incontinence; King's Health Questionnaire; Reliability; Validity
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is aimed to translate King's Health Questionnaire into Urdu language and to test its reliability and validity among Pakistani women with urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Having symptoms of Urinary Incontinence
* Age 21 or more than years
* Sufficient literacy to complete questionnaire

Exclusion Criteria:

* Being unable to complete questionnaires due to language and cognitive limitations
* Pelvic organ prolapse
* Concomitant neurological disorders

Ages: 21 Years to 83 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Females presenting with Urinary Incontinence
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-05-30 (Actual); Primary Completion 2022-07-25 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
King's Health Questionnaire | 7th day
  Change from Baseline (1st day)The King's Health Questionnaire is a disease-specific health-related quality-of-life instrument to measure health-related quality-of-life of patients with urinary incontinence

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Faisalabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No